CLINICAL TRIAL: NCT02213380
Title: Effect of Regional Anaesthesia and General Anaesthesia on Postoperative Delirium in Elderly Patients Undergoing Hip Fracture Surgery: a Multicenter Randomized Controlled Trial.
Brief Title: Effect of Anesthesia on Post-operative Delirium in Elderly Patients Undergoing Hip Fracture Surgery
Acronym: RAGADelirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Collaborators: National Research Institute for Family Planning, China (Other Government)
Responsible Party: Principal Investigator, Ting Li, associate chief physician, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RAGA-Delirium
Record Dates: First submitted 2014-08-05; First posted 2014-08-11 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Delirium
Keywords: delirium; general anesthesia; regional anesthesia; elderly patient; hip fracture
MeSH Terms: conditions — Emergence Delirium; Delirium; Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data collectors or outcome assessors, e.g. the medical staff who provide post-operative care in the ward and visit patients for preoperational assessment, hospital visits and subsequent follow-ups, will be blinded from group allocation throughout the study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group GA (Other): General anesthesia
  Interventions: Procedure: method of anesthesia
- group RA (Other): Regional anesthesia
  Interventions: Procedure: method of anesthesia

INTERVENTIONS:
Procedure: method of anesthesia — General anesthesia and regional anesthesia.
  General anesthesia(general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) will be used in group GA.
  Regional anesthesia(epidural, spinal, combined spinal and epidural anesthesia or nerve block) will be used in group RA

SUMMARY:
The purpose of this study is evaluate postoperative delirium after general anesthesia and regional anesthesia in elderly patients undergoing hip fracture surgery. Our research hypotheses are: (1) regional anesthesia may contribute to decrease the incidence of postoperative delirium. (2) Regional anesthesia may improve the outcome of elderly patient and reduce healthcare costs associated with postoperative delirium. (3) Postoperative delirium may result in poor long-term functional outcomes.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is an acute confusional state associated with changes in consciousness, arousal level and cognitive status. Elderly patients with hip fractures have the high incidence of delirium. The high risk factor of delirium include: Age 65 years or older, cognitive impairment/dementia, current hip fracture, severe illness and so on. Many previous studies predict that the majority of general anesthetic and sedative agents can favour postoperative delirium. However, none of studies have investigated the effect of general anesthesia and the effect of regional anesthesia and general anesthesia on the postoperative delirium in elderly patients undergoing hip fracture surgery in China. This multicentre, prospective, randomized controlled clinical trial is designed to evaluate postoperative delirium after general anesthesia and regional anesthesia in elderly patients undergoing hip fracture surgery. Our research hypotheses are: (1) regional anesthesia may contribute to decrease the incidence of postoperative delirium. (2) Regional anesthesia may improve the outcome of elderly patient and reduce healthcare costs associated with postoperative delirium. (3) Postoperative delirium may result in poor long-term functional outcomes.

This trial has the following nine investigational centers: Department of Anesthesiology, The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University, Wenzhou, China; Department of Anesthesiology, Tongji Hospital, Tongji Medical college, Huazhong University of Science & Technology, Wuhan, China; Department of Anesthesiology, West China Hospital of Sichuan University, Chengdu, China; Department of Anesthesiology, Southwest Hospital, Chongqing, China; Department of Anesthesiology, The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China; Department of Anesthesiology, Beijing Jishuitan Hospital, Beijing, China; Department of Anesthesiology, The First Affiliated Hospital of Nanchang University, Nanchang, China; Department of Anesthesiology, The Second Hospital of Anhui Medical University, Anhui, China; The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, China;

Eligible patients will be assigned into two study groups (group RA: regional anesthesia will be used, group GA: General anesthesia will be used) by centre-minimization randomization (web or telephone). There are 3 stratification factors: age (65-79,≥80), presence of delirium(yes, no), dementia(yes, no). There will be two teams of investigators involved in trial procedure and the patient's follow-up. Investigator A (experienced anesthetist), who are competent in caring for patients undergoing hip fracture surgery, will perform following works, which includes informed consent, randomization, anesthesia and recovery parameters. Investigator B will visit patient the day before surgery and 7days after surgery or until discharge to assess patient for presence, type and severity of delirium, collect other data during in hospital stay and follow up patients at 6 and 12 months. Investigator B will receive uniform training of using of CAM, Delirium Rating Scale-Revised-98 (DRS-R-98), MMSE and other test used in this trial) and will be not clear about protocol.

Within 24 h before surgery, cognitive function of each patient will be assessed with the MMSE, the presence of delirium will be diagnosed with the CAM, the type and severity of delirium will be assessed with DRS-R-98 and the pain will be assessed with a 100-mm visual analog scale (VAS). Routine monitoring (NBP, continuous ECG, and pulse oximetry) was initiated on all patients. Premedication for anesthesia will be avoided before surgery. Any medication impairing cognitive function will not be recommended, if administered, must be recorded it in detail.

Investigator A will allocated the patient into group GA or group RA according the centre-randomization with a unique registration number for each eligible patient. Treatment protocols for both groups will also stipulate no sedative be administrated during operation. Routine monitoring was initiated on all patients. Hypotension (Systolic Blood Pressure<90mmHg or drop of Mean Arterial Pressure>30%) should be treated with vasoactive agents or fluid boluses as deemed appropriate by anesthetists.

Postoperative analgesia will be administered according to the local procedures of each clinical trial site, aiming to maintain a VAS pain score ≤ 30 mm. Both groups will receive routine postoperative care on orthopedic ward.

All randomized patients will be followed up to 7 days after surgery (or discharge from the hospital). The 7 days follow-up includes: CAM, DRS-98-R (if applicable), VAS, Analgesic use (if applicable), Sedative use (if applicable), Post-operative morbidity and laboratory results (including serum hemoglobin, hematocrit, leucocytes, aspartate aminotransferase (AST), alanine aminotransferase (ALT), albumin, serum creatinine and urea concentrations, serum sodium and potassium and serum glucose concentration). Concomitant medications, adverse events and serious adverse events are record in all study visits. Economic parameters include: time to be discharged from post operation, total cost in hospital and cost for anesthesia of patient. Investigator B will also assess patient with POD in clinic or at their residence at 6 and 12 months to assess for presence of delirium, its type and severity (CAM, DRS-98-R), cognitive function using MMSE, and quality of life using The MOS 36-item Short-Form Health Survey (SF-36) questionnaire.

The study will be monitored regularly by the clinical research associate (CRA) through visits or telephone. CRA will verify the consistency of the data recorded on the case report forms with the source documents and the management of therapeutic batches, the presence and completeness of the investigator file.

ELIGIBILITY:
Inclusion Criteria:

* older patient (≥65 years)
* patient with hip fracture and planned hip fracture surgery
* patient willing to complete this study.

Exclusion Criteria:

* patient with multiple trauma or multiple fractures, pathological fractures, pelvic fractures, femur fractures
* contraindication (serious illness or medical conditions) for general anesthesia
* contraindication (infection at the site of needle insertion, coagulopathy, international normalized ratio >1.4, platelet count <80×109 litre-1, allergy to local anaesthetics and so on) for regional anesthesia;
* patient who cannot complete the preoperative mental tests (CAM and/or Mini-Mental State Examination (MMSE)) of this clinical trial
* patient known to susceptible to malignant hyperthermia
* known allergy or hypersensitivity to any drugs administered during this clinical trial
* previous participation in this clinical trial
* participation in another clinical trial within 4 weeks prior to selection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 950 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Gao, M.D., Study Chair — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Qingquan Lian, M.D., Study Chair — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Jun Li, M.D., Study Director — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Ting Li, M.D., Principal Investigator — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Joice Yeung, M.D., Study Director — Heart of England NHS Foundation Trust; Teresa Moledy, Study Director — Heart of England NHS Foundation Trust
Locations (13):
- China (13):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Tongji Hospital, Tongji Medical college, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The People's Hospital of Lishi, Lishi, Zhejiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Ningbo No.6 Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Jishuitan Hospital, Beijing
  - Southwest Hospital, Chongqing

REFERENCES:
- [Background] Sanders RD, Pandharipande PP, Davidson AJ, Ma D, Maze M. Anticipating and managing postoperative delirium and cognitive decline in adults. BMJ. 2011 Jul 20;343:d4331. doi: 10.1136/bmj.d4331. No abstract available. PMID 21775401
- [Background] Marcantonio ER, Flacker JM, Wright RJ, Resnick NM. Reducing delirium after hip fracture: a randomized trial. J Am Geriatr Soc. 2001 May;49(5):516-22. doi: 10.1046/j.1532-5415.2001.49108.x. PMID 11380742
- [Background] Bruce AJ, Ritchie CW, Blizard R, Lai R, Raven P. The incidence of delirium associated with orthopedic surgery: a meta-analytic review. Int Psychogeriatr. 2007 Apr;19(2):197-214. doi: 10.1017/S104161020600425X. Epub 2006 Sep 14. PMID 16973101
- [Background] Furlaneto ME, Garcez-Leme LE. Delirium in elderly individuals with hip fracture: causes, incidence, prevalence, and risk factors. Clinics (Sao Paulo). 2006 Feb;61(1):35-40. doi: 10.1590/s1807-59322006000100007. Epub 2006 Mar 10. PMID 16532223
- [Background] Nie H, Zhao B, Zhang YQ, Jiang YH, Yang YX. Pain and cognitive dysfunction are the risk factors of delirium in elderly hip fracture Chinese patients. Arch Gerontol Geriatr. 2012 Mar-Apr;54(2):e172-4. doi: 10.1016/j.archger.2011.09.012. Epub 2011 Oct 19. PMID 22014763
- [Background] Eeles EM, Hubbard RE, White SV, O'Mahony MS, Savva GM, Bayer AJ. Hospital use, institutionalisation and mortality associated with delirium. Age Ageing. 2010 Jul;39(4):470-5. doi: 10.1093/ageing/afq052. PMID 20554540
- [Background] Zakriya K, Sieber FE, Christmas C, Wenz JF Sr, Franckowiak S. Brief postoperative delirium in hip fracture patients affects functional outcome at three months. Anesth Analg. 2004 Jun;98(6):1798-1802. doi: 10.1213/01.ANE.0000117145.50236.90. PMID 15155351
- [Background] Kat MG, Vreeswijk R, de Jonghe JF, van der Ploeg T, van Gool WA, Eikelenboom P, Kalisvaart KJ. Long-term cognitive outcome of delirium in elderly hip surgery patients. A prospective matched controlled study over two and a half years. Dement Geriatr Cogn Disord. 2008;26(1):1-8. doi: 10.1159/000140611. Epub 2008 Jul 9. PMID 18562793
- [Background] Kat MG, de Jonghe JF, Vreeswijk R, van der Ploeg T, van Gool WA, Eikelenboom P, Kalisvaart KJ. Mortality associated with delirium after hip-surgery: a 2-year follow-up study. Age Ageing. 2011 May;40(3):312-8. doi: 10.1093/ageing/afr014. Epub 2011 Mar 17. PMID 21414946
- [Background] Fong TG, Jones RN, Shi P, Marcantonio ER, Yap L, Rudolph JL, Yang FM, Kiely DK, Inouye SK. Delirium accelerates cognitive decline in Alzheimer disease. Neurology. 2009 May 5;72(18):1570-5. doi: 10.1212/WNL.0b013e3181a4129a. PMID 19414723
- [Background] Witlox J, Slor CJ, Jansen RW, Kalisvaart KJ, van Stijn MF, Houdijk AP, Eikelenboom P, van Gool WA, de Jonghe JF. The neuropsychological sequelae of delirium in elderly patients with hip fracture three months after hospital discharge. Int Psychogeriatr. 2013 Sep;25(9):1521-31. doi: 10.1017/S1041610213000574. Epub 2013 May 7. PMID 23651760
- [Background] Cole MG. Persistent delirium in older hospital patients. Curr Opin Psychiatry. 2010 May;23(3):250-4. doi: 10.1097/YCO.0b013e32833861f6. PMID 20224406
- [Background] Young J, Murthy L, Westby M, Akunne A, O'Mahony R; Guideline Development Group. Diagnosis, prevention, and management of delirium: summary of NICE guidance. BMJ. 2010 Jul 28;341:c3704. doi: 10.1136/bmj.c3704. No abstract available. PMID 20667955
- [Background] Sanders RD. Hypothesis for the pathophysiology of delirium: role of baseline brain network connectivity and changes in inhibitory tone. Med Hypotheses. 2011 Jul;77(1):140-3. doi: 10.1016/j.mehy.2011.03.048. Epub 2011 Apr 16. PMID 21498007
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] Abou-Setta AM, Beaupre LA, Rashiq S, Dryden DM, Hamm MP, Sadowski CA, Menon MR, Majumdar SR, Wilson DM, Karkhaneh M, Mousavi SS, Wong K, Tjosvold L, Jones CA. Comparative effectiveness of pain management interventions for hip fracture: a systematic review. Ann Intern Med. 2011 Aug 16;155(4):234-45. doi: 10.7326/0003-4819-155-4-201108160-00346. PMID 21844549
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Huang MC, Lee CH, Lai YC, Kao YF, Lin HY, Chen CH. Chinese version of the Delirium Rating Scale-Revised-98: reliability and validity. Compr Psychiatry. 2009 Jan-Feb;50(1):81-5. doi: 10.1016/j.comppsych.2008.05.011. Epub 2008 Aug 23. PMID 19059519
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Derived] Li T, Li J, Yuan L, Wu J, Jiang C, Daniels J, Mehta RL, Wang M, Yeung J, Jackson T, Melody T, Jin S, Yao Y, Wu J, Chen J, Smith FG, Lian Q; RAGA Study Investigators. Effect of Regional vs General Anesthesia on Incidence of Postoperative Delirium in Older Patients Undergoing Hip Fracture Surgery: The RAGA Randomized Trial. JAMA. 2022 Jan 4;327(1):50-58. doi: 10.1001/jama.2021.22647. PMID 34928310
- [Derived] Li T, Yeung J, Li J, Zhang Y, Melody T, Gao Y, Wang Y, Lian Q, Gao F; RAGA-Delirium Investigators. Comparison of regional with general anaesthesia on postoperative delirium (RAGA-delirium) in the older patients undergoing hip fracture surgery: study protocol for a multicentre randomised controlled trial. BMJ Open. 2017 Oct 22;7(10):e016937. doi: 10.1136/bmjopen-2017-016937. PMID 29061612

RESULTS

PARTICIPANT FLOW:
Groups:
- Group RA: Regional anesthesia(epidural, spinal, combined spinal and epidural anesthesia or nerve block) will be used in group RA
- Group GA: General anesthesia (general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) will be used in group GA.
Period: Underwent Randomization
Arm/Group | Group RA | Group GA
Started | 476 | 474
Completed | 471 | 471
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Not treated | 3 | 3
Period: Per-protocol Analysis
Arm/Group | Group RA | Group GA
Started | 471 | 471
Completed | 439 | 435
Not Completed | 32 | 36
Not completed — Protocol Violation | 32 | 36

BASELINE CHARACTERISTICS:
Population: 950 patients were randomized and by intention-to-treat principal, 471 patients entered in to the RA group and 471 entered into the GA group.
Groups:
- Group GA: General anesthesia(general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) will be used in group GA.
- Total: Total of all reporting groups
Arm/Group | Group GA | Group RA | Total
Number analyzed (Participants) | 471 | 471 | 942
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.69 (6.57) | 77 (6.5) | 76.84 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 343 | 695
  Male | 119 | 128 | 247
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.79 (3.33) | 21.71 (3.48) | 21.75 (3.40)
Level of education [Count of Participants; unit: Participants]
  Illiterate | 282 | 286 | 568
  Elementary school | 119 | 124 | 243
  Secondary school or above | 70 | 61 | 131
Type of fracture [Count of Participants; unit: Participants]
  Femoral neck fracture | 264 | 278 | 542
  Fracture of femoral head | 1 | 2 | 3
  Intertrochanteric | 200 | 183 | 383
  Subtrochanteric | 6 | 8 | 14
ASA class [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) physical status classification system is a system for assessing the fitness of patients before surgery, the higher of the grade the worse.
  I A normal healthy patient II A patient with mild systemic disease III A patient with severe systemic disease IV A patient with severe systemic disease that is a constant threat to life.
  Participants
    I | 17 | 22 | 39
    II | 363 | 350 | 713
    III | 90 | 98 | 188
    IV | 1 | 1 | 2
Mini-mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills, and measured by scores range from zero [severe cognitive impairment] to 30 [normal cognition].
  units on a scale | 19.59 (6.41) | 19.39 (6.27) | 19.49 (6.34)
Pre-operative delirium [Count of Participants; unit: Participants] | 3 | 5 | 8
Comorbidities [Number; unit: participants]
  Respiratory system disease | 43 | 37 | 80
  Central nervous system disease | 57 | 65 | 122
  Urinary system disease | 117 | 112 | 229
  Gastrointestinal system disease | 145 | 173 | 318
  Hematologic system disease | 19 | 18 | 37
  Cardiovascular system disease | 300 | 280 | 580

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Delirium in 7 Days Post Operation
Description: Post-operative delirium diagnosed with Confusion Assessment Method
Time Frame: in 7 days post operation
Measure: Count of Participants; unit: Participants
Groups:
- Group RA: Method of anesthesia: regional anesthesia
  method of anesthesia: Method of anesthesia includes: general anesthesia and regional anesthesia.
  General anesthesia(general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) will be used in group GA.
  Regional anesthesia(epidural, spinal, combined spinal and epidural anesthesia or nerve block) will be used in group RA
- Group GA: Method of anesthesia: general anesthesia
  method of anesthesia: Method of anesthesia includes: general anesthesia and regional anesthesia.
  General anesthesia(general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) will be used in group GA.
  Regional anesthesia(epidural, spinal, combined spinal and epidural anesthesia or nerve block) will be used in group RA
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 471 | 470
Participants | 29 | 24

2. Secondary Outcome: Number of Participants With Post-operative Delirium
Description: Number of participants with delirium includes patients who had delirium in the post in the first 7 post-operative days.
  The severity of delirium was described using a severity score from 0 (no delirium) to 39 (highest severity) and subtypes of delirium as hyperactive, hypoactive or mixed.
Time Frame: within fist 7days post operation
Measure: Count of Participants; unit: Participants
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 29 | 24
Participants
  1 episode of POD | 16 | 10
  2 episodes of POD | 5 | 10
  >=3 episodes of POD | 8 | 4

3. Secondary Outcome: Severity of Delirium
Description: The worst severity scores of delirium was diagnosed with the DRS-R-98 within 7 days
Time Frame: within first 7days post operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 29 | 24
score on a scale | 23.48 (7.16) | 24.22 (7.04)

4. Secondary Outcome: The Subtypes of Delirium Diagnosed in 7 Days Post Operation
Description: The subtypes of delirium diagnosed with the Delirium Rating Scale-Revised-98 (DRS-R-98).
  Patients with the hyperactive subtype may be agitated, disoriented, and delusional, and may experience hallucinations. This presentation can be confused with that of schizophrenia, agitated dementia, or a psychotic disorder.
Time Frame: within first 7 days post operation
Measure: Count of Participants; unit: Participants
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 29 | 24
Participants
  Hyperactive | 16 | 16
  Hypoactive | 2 | 1
  Mixed motor | 2 | 3
  No motor | 9 | 4

5. Secondary Outcome: 30 Day Mortality
Description: Mortality within 30 days post operation
Time Frame: 30 days after surgery
Population: 6 patients in RA were lost to 30-day follow-up and 24 patients in GA were lost to 30-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 465 | 447
Participants | 8 | 4

6. Secondary Outcome: Acute Pain Score Using Visual Analogue Scale (VAS)
Description: The worst pain score within 7 days post-operation in both groups. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between no pain(0 point) to worst pain (100 points).
Time Frame: In 7days post operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 471 | 470
score on a scale | 0 [0 to 20] | 0 [0 to 10]

7. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay are measured from the anesthesia starting day to the discharge day
Time Frame: till the day of discharge from hospital, an average of 7 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 471 | 471
days | 7 [5 to 10] | 7 [6 to 10]

8. Secondary Outcome: Costs of Anesthetic Procedure
Description: Costs of anesthetic procedure only
Time Frame: 1 day after operation
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 471 | 471
dollars | 159 [110 to 220] | 268 [201 to 359]

9. Secondary Outcome: Total In-hospital Costs
Description: Entire expenditure in-hospital
Time Frame: till the day of discharge
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Group RA | Group GA
Number analyzed (Participants) | 471 | 471
dollars | 5582 [4598 to 7362] | 5908 [4778 to 7631]

10. Secondary Outcome: 6 Months Incidence of Delirium
Description: in clinic or at their residence, diagnosed with Confusion Assessment Method (CAM)
Time Frame: 6 months after discharge
Reporting Status: Not Posted, anticipated posting 2024-12

11. Secondary Outcome: 12 Months Incidence of Delirium
Description: in clinic or at their residence, diagnosed with Confusion Assessment Method (CAM)
Time Frame: 12 months after discharge
Reporting Status: Not Posted, anticipated posting 2024-12

12. Secondary Outcome: 6 Months Quality of Life
Description: using 36-Item Short Form Survey (SF-36) questionnaire
Time Frame: 6 months after discharge
Reporting Status: Not Posted, anticipated posting 2024-12

13. Secondary Outcome: 12 Months Quality of Life
Description: using 36-Item Short Form Survey (SF-36) questionnaire
Time Frame: 12months after discharge
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: Before discharge day with an average of 7 days, and for all cause mortality, is up to postoperative 30 days.
Arm/Group | Group RA | Group GA
All-Cause Mortality (participants affected / at risk) | 8/471 | 4/471
Serious Adverse Events (participants affected / at risk) | 3/471 | 2/471
Other Adverse Events (participants affected / at risk) | 83/471 | 79/471
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group RA (N=471) | Group GA (N=471)
acute myocardial infarction (Cardiac disorders) | 1 | 0
acute left heart failure (Cardiac disorders) | 1 | 0
acute gastric perforation (Gastrointestinal disorders) | 1 | 0
lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group RA (N=471) | Group GA (N=471)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Hypotension (Vascular disorders) | 13 | 10
Hypertension (Vascular disorders) | 4 | 13
Arrhythmia (Cardiac disorders) | 3 | 4
Chest distress (Cardiac disorders) | 3 | 2
Nausea and vomiting (Gastrointestinal disorders) | 47 | 34
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Acute gastric perforation* (Gastrointestinal disorders) | 1 | 0
Headache and dizziness (Nervous system disorders) | 2 | 4
Stroke (Nervous system disorders) | 0 | 1
Numbness in the back (General disorders) | 1 | 0
Shiver (General disorders) | 11 | 11
Pharyngodynia (General disorders) | 0 | 1
Skin allergy (Skin and subcutaneous tissue disorders) | 4 | 1
Mild burns of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Cerebrospinal fluid leak (Nervous system disorders) | 0 | 1
Hematoma in neck (General disorders) | 1 | 0
Hyperglycaemia (General disorders) | 0 | 1 — Hyperglycaemia (The elevated blood glucose is clinically significant compared to the baseline value, judged by the investigator)
Urinary retention (Renal and urinary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 — Anemia (myoglobin< 81g/L)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT02213380/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02213380/SAP_000.pdf